CLINICAL TRIAL: NCT03931551
Title: Effectiveness of Olaparib Plus Trastuzumab in HER2-positive BRCA-mutated Advanced Breast Cancer Patients (The OPHELIA Study)
Brief Title: Olaparib+Trastuzumab in HER2[+],Breast Cancer Susceptibility Gene (BRCA) Mutated Advanced Breast Cancer
Acronym: OPHELIA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Very slow recruitment due to subject profile
Sponsor: MedSIR (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP168; 2018-001213-32 (EudraCT Number)
Record Dates: First submitted 2019-04-17; First posted 2019-04-30 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2022-06

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — olaparib; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional Arm (Experimental): Olaparib tablet 300mg bd po + Herceptin (IV 4 mg/kg body followed by weekly doses of 2 mg/kg, or SC 600 mg every 3 weeks) until progression or unacceptable toxicity.
  Interventions: Drug: Olaparib [Lynparza®] plus Trastuzumab [Herceptin®]

INTERVENTIONS:
Drug: Olaparib [Lynparza®] plus Trastuzumab [Herceptin®] — Participants will receive olaparib (300 mg tablets, orally twice daily during 21-day cycles) in combination with herceptin (intravenous dose of 4 mg/kg body weight with subsequent weekly doses of 2 mg/kg or subcutaneous dose of 600 mg every 3 weeks) until progression or unacceptable toxicity.
  Other Names: Lynparza®; Herceptin®

SUMMARY:
This is a multicenter, open-label, single-arm, phase II clinical trial, phase II trial will evaluate the efficacy and safety of olaparib plus trastuzumab in patients with HER2[+], BRCA-mutated advanced breast cancer

DETAILED DESCRIPTION:
This open-label, multicenter, single arm, two cohorts, Simon's Two-Stage minimax design, phase II clinical trial will assess the efficacy of olaparib in combination with trastuzumab in patients with HER2-positive ABC with gene alterations in HRR DNA pathway. To be included in the cohort A of the study, patients must exhibit germinal deleterious mutations in BRCA1 or BRCA2 genes.

Eligible patients will have histologically proven diagnosis of adenocarcinoma of the breast with evidence of advanced disease, and at least one measurable disease as per RECIST v.1.1. Patients will have a documented history of progression on HER2-directed therapy for the treatment of HER2-positive breast cancer with not limits on prior therapies of chemotherapy and/or trastuzumab-lapatinib in advanced scenario, and at least one regimen of chemotherapy including trastuzumab.

The accrual goal will be a total of 20 patients

ELIGIBILITY:
Inclusion Criteria:

1. Obtention and signing of the molecular preselection consent regarding the mutational BRCA status confirmation prior to provision of the informed consent.
2. Provision of informed consent prior to any study specific procedures.
3. Male or female ≥18 years of age at the time of signing the Informed Consent Form (ICF).
4. Histologically and/or cytologically confirmed breast cancer with evidence of advanced disease (locoregionally recurrent or metastatic) not amenable to resection or radiation therapy with curative intent.
5. Patients with histologically and/or cytologically locally confirmed diagnosis of Human Epidermal Growth Factor Receptor 2 (HER2)-positive breast cancer according to the American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) May 2018 criteria.
6. Patients with documented germinal mutation in Breast Cancer (BRCA)1 or BRCA2 genes that is predicted to be deleterious or suspected deleterious (known or predicted to be detrimental/lead to loss of function). Patients with germinal BRCA1/2 mutations that are considered to be non-detrimental (e.g., "Variants of uncertain clinical significance" or "Variant of unknown significance" or "Variant, favor polymorphism" or "benign polymorphism," etc.) will not be eligible for the study. Patients with known germinal BRCA status prior to enrollment are considered eligible to participate.
7. Criteria of resistance to trastuzumab defined as:

   * Relapse on (neo) adjuvant treatment or within 6 months from completion, or
   * Progression on a trastuzumab regimen for advanced disease. No limitations on the number of prior trastuzumab regimens.
8. At least one prior systemic regimen for advanced disease including a pertuzumab or T-DM1 based regimen. No limitations on the number of prior systemic regimens.
9. Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 1.
10. Life expectancy greater or equal to 16 weeks.
11. Patients must have evaluable or measurable disease by Computed Tomography (CT) scan or Magnetic resonance imaging (MRI), according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
12. Patients must have normal organ and bone marrow function within 35 days prior to administration of study treatment as defined below:

    * Hematological: White blood cell (WBC) count >3.0 x 109/L, absolute neutrophil count (ANC) ≥1.5 x 109/L, platelet count ≥100.0 x109/L, and hemoglobin ≥ 10 g/dL
    * Hepatic: bilirubin ≤ 1.5 times the upper limit of normal (x ULN) (≤2.0 in patients with known Gilberts syndrome) or direct bilirubin ≤ 1 x ULN; alkaline phosphatase (ALP), Aspartate aminotransferase (AST) / Serum Glutamic Oxaloacetic Transaminase (SGOT), and Alanine aminotransferase (ALT) / Serum Glutamic Pyruvate Transaminase (SGPT) ≤ 2.5 x institutional ULN unless liver metastases are present, in which case they must be ≤ 5 x ULN.
    * Renal: Serum creatinine ≤ 1.5 x ULN or based on a 24-hour urine test or estimated creatinine clearance ≥ 51 mL/min using the Cockcroft-Gault equation:

    Estimated creatinine clearance = (140-age [years]) x weight (kg) (x F)a serum creatinine (mg/dL) x 72a where F=0.85 for females and F=1 for males.
13. Patients have been informed about the nature of study, including the exploratory studies and has agreed to participate and signed the ICF prior to participation in any study-related activities.
14. Males, postmenopausal and premenopausal women. Premenopausal women of childbearing potential (not undergoing to tubal ligation or hysterectomy) must have a negative blood or urine pregnancy test within 28 days prior to the start of study treatment and confirmed on Day 1 prior to commencing treatment

    * Postmenopausal status is defined as either:
    * Prior bilateral oophorectomy; Or
    * Age > 60 years; Or Age < 60 years and amenorrhoeic for 12 months in the absence of chemotherapy, tamoxifen, toremifene or ovarian suppression, and Follicle-stimulating hormone (FSH) and estradiol in postmenopausal range; Or Age < 60 years and taking tamoxifen or toremifene and FSH and plasma estradiol level in postmenopausal ranges; Or Radiation-induced castration with >1-year interval since last menses. Premenopausal status is defined as all those women who do not meet any of above criteria.

    Note: Documented hysterectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the patient must be willing to use 2 highly effective forms of contraception in combination male condom plus an acceptable hormonal or non-hormonal method) throughout the study. Information must be captured appropriately within the site's source documents. Correct forms of contraception for males and females are detailed in Appendix 5: Acceptable birth control methods.
15. Patients is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
16. Snap frozen or formalin fixed paraffin-embedded (FFPE) tumor sample is mandatory for exploratory central testing.
17. Patients must fulfil the relative field on the informed consent for donating blood samples and serial biopsies at baseline and on disease progression for the exploratory biomarker studies.

Exclusion Criteria:

1. Patients that have previously received any poly(ADP-ribose) polymerase (PARP) inhibitor (PARPi) for any reason, including olaparib.
2. Involvement in the planning and/or conduct of the study (applies to both Sponsor's staff and/or staff at the study site).
3. Patients simultaneously enrolled in any interventional clinical trial.
4. Patients who have received any systemic chemotherapy during the last 3 weeks prior initiating protocol therapy.
5. Patients who have had radiation therapy encompassing >20% of the bone marrow within 3 weeks prior to start of treatment, excepting for palliative radiation therapy to a small field >1-week prior to Day 1 of study.
6. Resting electrocardiogram (ECG) indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
7. Concomitant use of known strong Cytochrome P450 (CYP)3A inhibitors (e.g., itraconazole, telithromycin, clarithromycin, boosted protease inhibitors, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
8. Concomitant use of known strong (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil). The required washout period prior to starting study treatment is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
9. Persistent toxicities (Common Terminology Criteria for Adverse Events (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia.
10. Patients with Myelodysplastic syndrome (MDS) / Acute myeloid leukemia (AML) or with features suggestive of MDS/AML.
11. Patients having diagnosis, detection, or treatment of another type of cancer during the last 5 years prior to initiating protocol therapy (except adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, definitively treated ductal carcinoma in situ, stage 1, grade 1 endometrial carcinoma), or other solid tumors including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for ≤5 years).
12. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
13. Patients considered a high medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 6 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution CT scan or any psychiatric disorder that prohibits obtaining informed consent.
14. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
15. Immunocompromised patients (e.g., patients who are known to be serologically positive for human immunodeficiency virus and those with undetectable viral load).
16. Patients with a known hypersensitivity to olaparib or trastuzumab or any of the excipients of the products.
17. Clinically significant cardiovascular disease (stroke, unstable angina pectoris, or documented myocardial infarction) within 6 months prior to study entry; history of documented congestive heart failure (New York Heart Association II-III-IV); symptomatic pericarditis; documented cardiomyopathy; ventricular arrhythmias with the exception of benign premature ventricular contractions; conduction abnormality requiring a pacemaker; other arrhythmias not controlled with medication].
18. Left ventricular ejection fraction below 55% as determined by multiple-gated acquisition (MUGA) scan or echocardiography (ECHO).
19. Uncontrolled hypertension (systolic > 150 mm Hg and/or diastolic > 100 mm Hg) despite adequate antihypertensive treatment.
20. Patients currently receiving anti-coagulant therapy (low molecular weight heparin and warfarin with careful monitoring of patients are permitted), or another immunosuppressive agent (standard premedication for chemotherapy and local applications are allowed).
21. Patients with pulmonary disease requiring continuous oxygen therapy.
22. Previous history of bleeding diathesis.
23. Patients with known active hepatitis (i.e. Hepatitis B or C).
24. Patients with moderate or severe hepatic impairment.
25. Chronic daily treatment with corticosteroids with a dose of ≥ 10 mg/day methylprednisolone equivalent (excluding inhaled steroids), except for prophylaxis use.
26. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation.
27. Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment and in a dose < 10 mg/day methylprednisolone equivalent. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.

Female patients who are pregnant or breastfeeding, or adults of reproductive potential who are not using effective birth control methods.

Patients unwilling to or unable to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of olaparib in combination with trastuzumab | Baseline up to 12 months.
  as determined by the Clinical benefit rate (CBR) response (PR) divided by the number of patients in the analysis set- in patients with germinal BRCA-mutated [cohort A] based on local investigator's assessment according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria guidelines v.1.1.

SECONDARY OUTCOMES:
ORR | Baseline up to 30 months.
  ORR -defined as the number of patients with CR and PR divided by the number of patients in the analysis set- in patients with wild-type germinal BRCA/HRD-positive tumors [cohort B] based on local investigator's assessment according to RECIST criteria guidelines v.1.1.
PFS i | Baseline up to 30 months.
  PFS -defined as the period of time from treatment initiation to the first occurrence of disease progression or death from any cause, whichever occurs first- in patients with wild-type germinal BRCA/HRD-positive tumors [cohort B] based on local investigator's assessment according to RECIST criteria guidelines v.1.1.
Clinical benefit rate (CBR | Baseline up to 30 months.
  CBR -defined as the number of patients with CR, PR or stable disease (SD) divided by the number of patients in the analysis set- both in patients with germinal BRCA-mutated [cohort A] and wild-type germinal BRCA/HRD-positive [cohort B] tumors based on local investigator's assessment according to RECIST criteria guidelines v.1.1.
Duration of response (DoR) | From documented objective response up to 30 months.
  DoR -defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first- both in patients with germinal BRCA-mutated [cohort A] and wild-type germinal BRCA/HRD-positive [cohort B] tumors based on local investigator's assessment according to RECIST criteria guidelines v.1.1.
Maximum Tumor Shrinkage | Baseline up to 30 months.
  Maximum Tumor Shrinkage -defined as the percentage of tumor shrinkage from baseline [obtained from the sum of the largest diameters of the target lesions]- both in patients with germinal BRCA-mutated [cohort A] and wild-type germinal BRCA/HRD-positive [cohort B] tumors based on local investigator's assessment according to RECIST criteria guidelines v.1.1.
Overall survival (OS) | Baseline up to 30 months.
  OS -defined as the period of time from treatment initiation to death from any cause- both in patients with germinal BRCA-mutated [cohort A] and wild-type germinal BRCA/HRD-positive [cohort B] tumors based on local investigator's assessment according to RECIST criteria guidelines v.1.1.
Health-Related Quality of Life (HRQoL) in cohorts A and B | Baseline up to 30 months.
  Change from baseline in scores using the European Organisation for Research and Treatment of Cancer QoL Questionnaire Core 30 (QLQ-C30) [with 5 functional and 3 symptom scales, a Global Health Status (GHS)/QoL scale, and 6 single items], QLQ-BR23 [with 4 functional and 4 symptom scales], and EQ-5D [with 5 dimensions and a health status rating scales] modules at baseline, Day 1 of cycles 2-4, then on Day 1 of each subsequent cycle starting with cycle 6, and at the end-of-treatment. Responses to all items are converted to a 0-100 scale using a standard scoring algorithm. For functional scales, higher score represents a better level of functioning; for symptom scales, a higher score represents a higher severity of symptoms.
Safety adverse events (AEs) | Baseline up to 30 months.
  Number of patients with treatment-related AEs (Grade 3 and 4 AEs and serious adverse events [SAEs]) by using the National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) v.5.0.

OTHER OUTCOMES:
Exploratory Objective (prevalence of BRCA alterations) | Baseline up to 30 months.
  The number of patients with HER2[+], germinal BRCA1/2 mutated advanced breast cancer divided by the number of patients in the analysis set.
Exploratory Objective (predictive value of BRCA alterations) | Baseline up to 30 months.
  The number of patients with HER2[+], germinal BRCA1/2 mutated ABC who obtain best response, in terms of CR, PR, SD, or progressive disease (PD) divided by the number of patients in the analysis set.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Enrique Alés-Martínez, Principal Investigator — Complejo Hospitalario de Ávila
Locations (4):
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Clínico San Carlos, Madrid
  - Hospital Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: No
It is not planned